CLINICAL TRIAL: NCT00624377
Title: Safety and Effectiveness of Spiriva® in COPD (Chronic Obstructive Pulmonary Disease) Patients Under the Real Condition of Usual Practice
Brief Title: Safety and Effectiveness of Spiriva in COPD (Chronic Obstructive Pulmonary Disease) Patients Under the Real Condition of Usual Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.399
Record Dates: First submitted 2008-02-19; First posted 2008-02-27 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD patients
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — Tiotropium 18 mcg HandiHaler once daily

SUMMARY:
The purpose of this study is to monitor the change in the health status of severe COPD patients after the initiation of Tiotropium therapy. This will be assessed by the physician's global evaluation of the patient's health status on a 8-point scale. This measure has been shown to correlate with a established standard measure of the patients health related quality of life. The primary analysis in this trial will only include patients not pre-treated with a long-acting beta-agonist to establish a clear efficacy signal in this patient population. As the reality of COPD treatment nowadays is poly-pharmacy, a secondary analysis will analyse patients who are pretreated with long-acting bronchodilators to put the changes in the health status in a likely real world context. In parallel to these evaluations of the health status, the lung function response of the patients will be assessed to gain an established objective measure of treatment response.

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD; updated 2005).
2. Patients who are assessed to benefit from the intake of long-acting anticholinergics as a monotherapy or as add-on medication.
3. Tiotropium bromide naïve patients.
4. Patients with indication for tiotropium bromide according to Taiwanese Spiriva® label.

Exclusion criteria:

1. Patients with contraindications to tiotropium bromide use (as per the Spiriva® package insert).
2. Known hypersensitivity to the active ingredient or to any of the excipients of Spiriva®.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Probability Sample
Enrollment: 2031 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- Taiwan (16):
  - Boehringer Ingelheim Investigational Site, Chan Wha
  - Boehringer Ingelheim Investigational Site, Chiayi City
  - Boehringer Ingelheim Investigational Site, Hwa Lian
  - Boehringer Ingelheim Investigational Site 1, Kaohsiung City
  - Boehringer Ingelheim Investigational Site 2, Kaohsiung City
  - Boehringer Ingelheim Investigational Site 3, Kaohsiung City
  - Boehringer Ingelheim Investigational Site 1, Taichung
  - Boehringer Ingelheim Investigational Site 2, Taichung
  - Boehringer Ingelheim Investigational Site, Tainan
  - Boehringer Ingelheim Investigational Site 1, Taipiei
  - Boehringer Ingelheim Investigational Site 2, Taipiei
  - Boehringer Ingelheim Investigational Site 3, Taipiei
  - Boehringer Ingelheim Investigational Site 4, Taipiei
  - Boehringer Ingelheim Investigational Site 5, Taipiei
  - Boehringer Ingelheim Investigational Site 6, Taipiei
  - Boehringer Ingelheim Investigational Site, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2,031 patients were enrolled between Jan-11-2008 to Mar-24-2010
Period: Overall Study
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Started | 2031
Completed | 1387
Not Completed | 644
Not completed — Lost to Follow-up | 355
Not completed — Withdrawal by Subject | 100
Not completed — Adverse Event | 14
Not completed — Other | 91
Not completed — Non-evaluable population | 84

BASELINE CHARACTERISTICS:
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 2031
Age, Customized [Mean (Standard Deviation); unit: Year] — The number is different than the overall number of baseline participants because some of the CRF have lost during the follow up of the patient.
  Year | 72.87 (10.32)
Gender [Number; unit: Participants] — The number is different than the overall number of baseline participants because some of the CRF have lost during the follow up of the patient.
  Participants
    Female | 245
    Male | 1781
Weight [Mean (Standard Deviation); unit: kg] — The number is different than the overall number of baseline participants because some of the CRF have lost during the follow up of the patient.
  kg | 61.94 (11.60)
Height [Mean (Standard Deviation); unit: cm] — The number is different than the overall number of baseline participants because some of the CRF have lost during the follow up of the patient.
  cm | 162.57 (7.38)

OUTCOME MEASURES:

1. Primary Outcome: Change of Physician's Global COPD (Chronic Obstructive Pulmonary Disease) Assessment After 8-week of Treatment Severe COPD Patients Without Concomitant LABA (Long-acting Beta Agonists) Treatment
Description: The extent of satisfaction with tiotropium bromide treatment was evaluated based on the changes of the Global COPD Assessment performed by the physician. This evaluation was done with the help of an 8-point scale rated from 1 (Poor) to 8 (Excellent) following the question "Overall, how is the COPD of your patient?"
Time Frame: Baseline and 8 weeks
Population: Safety population:
  Safety population will be defined as all patients enrolled in the study. Safety endpoints will be analyzed based on the safety population.
  Complete population:
  Complete population was defined as the subjects who completed 3 visit measurements. Efficacy endpoints will be analyzed based on the completed population.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 232
Units on a Scale | 1.16 (1.34)

2. Primary Outcome: Changes of FEV1 (Forced Expiratory Volume In 1 Second) After 8 Weeks of Treatment
Description: FEV1: Average values for FEV1 in healthy people depend mainly on sex and age. Values of between 80% and 120% of the average value is considered normal. FEV1 < 80% of the predicted value in combination with an FEV1/FVC < 70% confirms the presence of airflow limitation that is not fully reversible
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter per second
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 1386
liter per second | 6.27 (12.99)

3. Primary Outcome: Changes of FEV1/FVC (Forced Vital Capacity) After 8 Weeks of Treatment
Description: FEV1/FVC (FEV1%) is the ratio of FEV1 to FVC. In healthy adults this should be approximately 75-80%. In obstructive diseases, the value often decreased (<80%, often ~45%).
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 1383
Ratio | 4.36 (10.72)

4. Secondary Outcome: Change of Physician's Global COPD Assessment (8-point Scale) After 8-week of Treatment in Severe COPD Patients Independent of Concomitant LABA Treatment
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 408
Units on a Scale | 1.72 (1.77)

5. Secondary Outcome: Change of Physician's Global COPD Assessment (8-point Scale) After 8-week of Treatment in All COPD Patients Without Concomitant LABA Treatment
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 913
Units on a Scale | 1.19 (1.31)

6. Secondary Outcome: Change of Physician's Global COPD Assessment (8-point Scale) After 8-week of Treatment in All COPD Patients Independent of Concomitant LABA Treatment
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 1387
Units on a Scale | 1.54 (1.67)

7. Secondary Outcome: Change of Patient's Global COPD Assessment (8-point Scale) After 8-week of Treatment Grouped According to Patients Severity and Concomitant Medication With LABAs
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 247
Units on a Scale | 2.84 (2.21)

8. Secondary Outcome: Percentage of Participants Which Had a Reduction of Concomitant Drug Use
Description: The Physician has been asked to record any prescribed and other medication used for COPD (at the physician discretion) at every visit.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Number analyzed (Participants) | 1387
Percentage of Participants | 76

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Spiriva 18µg With HandiHaler Device on COPD Patients
Serious Adverse Events (participants affected / at risk) | 16/2031
Other Adverse Events (participants affected / at risk) | 0/2031
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva 18µg With HandiHaler Device on COPD Patients (N=2031)
Cardiac disorder (Cardiac disorders) | 1
Death (General disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory therapy (Surgical and medical procedures) | 1
Infarction (Vascular disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 2
Cynosis (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.